CLINICAL TRIAL: NCT02518997
Title: Effects of Reading to Preterm Infants on Baby and Parents' Well Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Melissa Scala, Assistant Professor of Pediatrics, Georgetown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-1464
Record Dates: First submitted 2015-03-10; First posted 2015-08-10 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Parental Infant Bonding; Cardio-respiratory Stability in Preterm NICU Infants
Keywords: Preterm Infants; Bedside Reading aloud; Parental wellbeing; Parental Bonding; cardio-respiratory stability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All enrolled infants (Experimental): All participants will have Parental Reading Aloud at the prescribed intervals while being monitored for cardio-respiratory stability.
  Interventions: Other: Parental Reading Aloud

INTERVENTIONS:
Other: Parental Reading Aloud — Infants will be exposed to parental reading aloud or to a recording of the parent's voice reading during times of cardio-respiratory monitoring.

SUMMARY:
Reading to children is believed to be beneficial to cognitive and mental development.This study will examine the response of premature Neonatal Intensive Care Unit (NICU) infants to bedside reading by measuring changes in heart rate, blood pressure, breathing and oxygen levels. The investigators will follow rates of common preterm health issues while in the hospital and time to hospital discharge. Effects of bedside reading on parental stress and infant bonding will be measured and compared to usual rates of these indicators to determine if reading to babies reduces stress and enhances bonding.

DETAILED DESCRIPTION:
The NICU at Georgetown University Hospital cares for approximately 100 infants per year in the study population between 26-34 weeks gestation. We have a patient population where parental daily visits are the norm, allowing for a study using live voices.

The investigators will approach parents of infants who meet entry criteria who are nearing one week of age after consultation with the clinical care team to determine stability. All preterm infants admitted to the NICU who are deemed stable enough to participate by the primary team will be approached for study participation.

After parental consent is obtained, the parents will be given an initial questionnaire to assess demographic data such as parental education and attitudes regarding reading to infants. Parents will be given a picture book with rhythmic sound patterns for reading aloud to their infant. Bedside nurses will help guide parents to the best time for infant reading. Time of parent reading (start and stop time) will be recorded in the infant's chart. Mothers and fathers will be allowed to read to the infant at separate reading times. A decibel monitor placed at the opening of the incubator will display the decibel level of parental voice.

Parents will be asked to read to their babies for at least 15 minutes but not more than 60 minutes per session. The total reading time for any 24 hour period can be up to 90 minutes.

Reading will occur with the infant in an incubator, in an open warmer or crib or while being held by parents. If the infant is in an incubator, parents will read with the portal closest to the parent open. For those babies who are in an open crib or warmer the parents will read close enough to the bedside so as not to be heard by neighboring patients. In older infants who are stable enough for kangaroo care or are out of bed being held by parents, reading can occur at those times, if desired by the parents. The Infant's location (in incubator, open bed, kangaroo care or parental holding) will be recorded in a study bedside binder.

Parents may also make a 30 minute recording on a digital recording device which can be played back to the baby twice per day if the parents are not expected to visit and the total reading time has not been met. Nursing staff will alternate between mother and father recorded sessions when neither parent is present and the total reading time for the day has not occurred.

Enrolling 80 infant/parent pairs will allow for subgroup analysis of Cardio Respiratory Events (CREs) in different corrected gestational ages (grouped into two cohorts 26-30 completed weeks and 31-34 completed weeks) and for comparison in effect of maternal and paternal voices. The study will not dictate who reads when both parents are present, but will encourage fathers to read if their visits are less frequent than mother's.

To assess changes in CREs, during NICU admission we will continuously record infant heart rate, respiratory rate, oxygen saturation, and CREs via software capable of downloading data directly from infant monitors used for routine clinical monitoring in the NICU, reducing variations in bedside charting and supplying a more complete documentation of the infant's cardiopulmonary status. Assessment of parental reading impact will be assessed at least three times per week and up to twice per day. Monitoring equipment is limited to recording three infants at one time so number of infants monitored per day will be impacted by total number of infants in the study at one time.

Changes in heart rate, respiratory rate, numbers of desaturation and apnea or bradycardia events will be scored for 3 reading session epochs; one hour before reading, during reading and one hour after parent reading will be measured. We will also compare CRE scores of reading times to CRE scores of similar periods throughout the day (eg 30 minutes before and after feedings). Enrolled infants who require high frequency ventilation will be temporarily withdrawn until the infant returns to conventional ventilation. If an infant is deemed too ill to participate by the primary team due to worsening in clinical status, he or she may be temporarily withdrawn until the primary team decides he/she is again stable enough to participate.

Parent-infant bonding will be assessed via a questionnaire administered four times during the study: before enrollment, at hospital discharge (average expected length of time 6 weeks) and 3-months after discharge. Attitudes toward reading to infants and patterns of reading at home after discharge will also be recorded and compared.

Frequency of parent-infant reading after discharge will be compared to historical controls via survey of families whose infants have been discharged from the NICU prior to the study initiation and exposure to subsequent study-initiated reading education efforts. This control group will be polled for parental education, feelings on reading to infants and frequency of that behavior at home in the first 3 months after hospital discharge to obtain a historical baseline for our study population. Parents of the prospective reading group will receive the same questionnaire at 3 months after discharge and these results will be compared.

Data on CREs will be recorded at multiple time points for the duration of care within an incubator and outcomes followed to hospital discharge, an average of 8 weeks. Parent-infant reading patterns will be followed up to 3 months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Infants between 26 0/7 34 6/7 weeks corrected gestational age (CGA) at the time of enrollment, [gestational age stated as # of weeks plus the number of days of the next week completed, the days are expressed as a fraction of a 7 day week (CGA= GA at birth + days of life)] rationale: 26 0/7 is the age at which the auditory system is generally well formed but still immature. Infants born at less than 26 0/7 weeks GA can be enrolled once they reach 26 0/7 weeks.
2. Infants at least 7 days of life to allow for transition to extrauterine life.

Parental Inclusion Criteria

1. Agreement to the study with signed Informed Consent Form and HIPAA Authorization
2. Visits on a regular basis (at least 3 times per week)
3. Is literate (able to read)

Exclusion Criteria:

1. Infants deemed too ill to participate by the primary care team at one week of age, although those infants may be enrolled at a later date when they are stabilized with the approval of the clinical care team,
2. infants with congenital hearing loss,
3. chromosomal abnormalities,
4. infants not expected to survive.

Parents Exclusions Does not read or is uncomfortable reading aloud. (unlikely to sign informed consent if this is the case)

-

Ages: 7 Days to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2014-10; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Scala, MD, Principal Investigator — Georgetown University
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Enrolled Infants
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Infants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: days] | 27.8 [8 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18
gestational age at birth [Mean (Full Range); unit: weeks] | 25.8 [23 to 31]
postmenstrual age at study entry [Mean (Full Range); unit: weeks] | 30 [26 to 34]
Birth weight [Mean (Full Range); unit: grams] | 831 [540 to 1430]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Oxygen Saturation Measurements <85%
Description: Percent of measured oxygen saturations recorded as less than 85%
Time Frame: While the infant is hospitalized, equipment is available and cared for in an incubator, an average of 2-6 weeks
Population: All enrolled infants had measured oxygen saturations at 4 time periods: during reading exposure and 3 hours before reading, 1 hour before reading and 1 hour after reading
Measure: Mean (Full Range); unit: Percent Oxygen saturation measurements
Units Other Than Participants: Oxygen saturation measurements
Groups:
- All Enrolled Infants: Infants exposed to parental reading-all enrolled infants
- Infants 3 Hours Before Reading: Infants with oxygen saturations measured 3 hours before reading exposure
  All enrolled infants
- Infants 1 Hour Before Reading Exposure: All enrolled infants. Infants with oxygen saturations measured 1 hour before reading exposure
- Infants 1 Hour After Reading Exposure: Infants with oxygen saturation data measured 1 hour after reading exposure
  All enrolled infants
Arm/Group | All Enrolled Infants | Infants 3 Hours Before Reading | Infants 1 Hour Before Reading Exposure | Infants 1 Hour After Reading Exposure
Number analyzed (Participants) | 18 | 18 | 18 | 18
Number analyzed (Oxygen saturation measurements) | 23986 | 23921 | 23030 | 23198
Percent Oxygen saturation measurements | 15.2 [0 to 62.1] | 16.94 [0 to 70.9] | 17.65 [0 to 64.6] | 14.39 [0 to 87.0]

ADVERSE EVENTS:
Time Frame: For the extent of the infant's hospitalization, up to 6 months
Arm/Group | All Enrolled Infants
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
The number of reading events at the lowest gestational ages was limited and an equal number of reading events were unavailable for all infants at all gestational ages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02518997/Prot_SAP_000.pdf